CLINICAL TRIAL: NCT06841406
Title: Budesonide as a Treatment for Low-grade Duodenal Inflammation in Functional Dyspepsia
Brief Title: Budesonide as a Treatment for Functional Dyspepsia
Acronym: BuDy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S64291
Record Dates: First submitted 2025-02-11; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2024-12

CONDITIONS: Functional Dyspepsia
Keywords: Functional Dyspepsia; Budesonide; Low-grade immune activation; Eosinophils; Mast cells; Postprandial distress syndrome; Disease; Pathologic Processes; Gastrointestinal Diseases; Gastrointestinal Diseases, Functional; Digestive System Diseases
MeSH Terms: conditions — Disease; Pathologic Processes; Gastrointestinal Diseases; Digestive System Diseases | interventions — Budesonide; Mannitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Budesonide, 9mg, oral use (Experimental): Budesonide, 9mg, oral use, once daily, 30 minutes before meal
  Interventions: Drug: budesonide
- Mannitol, 9mg, oral use (Placebo Comparator): Mannitol, 9mg, oral use, once daily, 30 minutes before meal
  Interventions: Drug: Mannitol

INTERVENTIONS:
Drug: budesonide — During an 8-week treatment period, patients will receive 9 mg of Budesonide daily, administered orally in enteric-coated capsules. Following this period, participants will undergo a gradual dose reduction to minimize the risk of adrenal insufficiency: 6 mg daily for 2 weeks, followed by 3 mg daily for another 2 weeks before discontinuing treatment.
  Arms: Budesonide, 9mg, oral use
Drug: Mannitol — During an 8-week treatment period, patients will receive 9 mg of Mannitol daily, administered orally in enteric-coated capsules as placebo control. Following this period, participants will undergo a gradual dose reduction as is the case in the experimental group: 6 mg daily for 2 weeks, followed by 3 mg daily for another 2 weeks before discontinuing treatment.
  Arms: Mannitol, 9mg, oral use

SUMMARY:
This clinical study is being conducted to evaluate the investigational drug, Budesonide, for the treatment of functional dyspepsia. The goal of this study is to learn more about the effect of Budesonide on patients with functional dyspepsia. Budesonide is a well-known and commonly used drug, and is part of the recommended therapy for patients with inflammatory bowel diseases (Crohn's disease or ulcerative colitis). It is also used as inhalation therapy for respiratory conditions such as asthma and COPD. However, the effect of Budesonide in patients with functional dyspepsia is still unknown. In patients with functional dyspepsia, an increased presence of inflammatory cells has been observed in the duodenum. Budesonide may reduce inflammatory responses.

Therefore, with this study, the investigators aim to investigate primarily:

1. Whether Budesonide has an effect on the inflammatory cells observed in functional dyspepsia.
2. Whether the symptoms of patients with functional dyspepsia improve during and after taking Budesonide.
3. Whether inflammatory cells could be the cause of symptoms in functional dyspepsia.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Functional dyspepsia (subtype postprandial distress syndrome) as per Rome IV diagnostic criteria

   * Symptom characteristics of dyspepsia (upper gastrointestinal symptoms occurring in the last 3 months and meal related)
   * Negative endoscopy (maximum 12 months old)
2. Patients must provide witnessed written informed consent prior to any study procedures being performed
3. Patients aged between 18 and 70 years inclusive
4. Male or female patients
5. Women of child-bearing potential agree to apply a highly effective method of birth control during the entire duration of the trial. Highly effective birth control is defined as those which result in a low failure rate (i.e., less than 1% per year) when used constantly and correctly such as implants, injectables, combined oral contraceptive method, or some intrauterine devices (IUDs), sexual abstinence, or vasectomized partner. Women of non-childbearing potential may be included if surgically sterile (tubal ligation or hysterectomy) or postmenopausal with at least 2 year without spontaneous menses
6. Subjects who are capable to understand the study and the questionnaires, and to comply with the study requirements

Exclusion Criteria:

1. Patients with any condition which, in the opinion of the investigator, makes the patient unsuitable for entry into the study
2. Patients with any major psychiatric disorders (including those with a major psychosomatic element to their gastrointestinal disease), depression, alcohol or substance abuse in the last 2 years
3. Patients presenting with predominant symptoms of irritable bowel syndrome (IBS) or of gastro-esophageal reflux disease (GERD)
4. Presence of diabetes mellitus, celiac disease (diagnosed with presence of anti-tissue transglutaminase antibodies and anti-gliadin antibodies or via duodenal biopsies), lupus, scleroderma or other systemic auto-immune disease
5. Patients with eosinophilic esophagitis or eosinophilic gastroenteritis
6. Active H. Pylori infection (or < 6 months after eradication)
7. Organic gastro-intestinal disease of history of gastrointestinal surgery other than appendectomy
8. Known impaired liver dysfunction
9. Drugs altering gastric emptying, anti-inflammatory drugs, acid suppressive drugs or some drugs altering the CYP3A4 metabolism
10. Major change in diet last 3 months
11. Females who are pregnant or lactating
12. Patients not capable to understand or be compliant with the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Effect of Budesonide on the reduction of the number of eosinophils on duodenal biopsies in patients with functional dyspepsia | before treatment and 8 weeks after start of treatment (9 mg)
  The primary endpoint is to evaluate the effect of Budesonide on duodenal eosinophilia (30% reduction) in patients with functional dyspepsia.

SECONDARY OUTCOMES:
The effect of budesonide in functional dyspepsia on gastric emptying time. | before treatment and 8 weeks after start of treatment (9 mg)
  The effect of budesonide in functional dyspepsia on gastric emptying time, assessed by 13C-octanoic acid gastric emptying breath test
The effect of budesonide in functional dyspepsia on symptom outcome using the Leuven Postprandial Distress Scale (range 0-4; 0 = no symptoms, 4 = very severe symptoms) | Daily for 2 weeks before start of treatment. Daily during the 8 weeks of treatment (at 9 mg). Daily during the 4 weeks of tapering the treatment
  The effect of budesonide in functional dyspepsia on gastro-intestinal symptoms of patients, based on the Leuven Postprandial Distress Scale (LPDS, range 0-4; 0 = no symptoms, 4 = very severe symptoms)
The effect of budesonide in functional dyspepsia on Quality of life of patients | At baseline, 8 weeks after start of treatment (9mg), 2 weeks after start of tapering (which is at 10 weeks), at the end of tapering (at 12 weeks), at 16 weeks (4 weeks after treatment discontinuation)
  Effect of Budesonide on the Impact of Functional Dyspepsia Symptoms on Patients' Quality of Life, Assessed by the 30-Item PAGI-QoL Questionnaire (Likert Scale 0-5; 0 = No Impact, 5 = Constant Impact)
The effect of budesonide in functional dyspepsia on Quality of life of patients | At baseline, 8 weeks after start of treatment (9mg), 2 weeks after start of tapering (which is at 10 weeks), at the end of tapering (at 12 weeks), at 16 weeks (4 weeks after treatment discontinuation)
  Effect of Budesonide on the Impact of Functional Dyspepsia Symptoms on Patients' Quality of Life, Assessed by the SF-NDI Questionnaire (10 items, covering five domains; Likert Scale 0-5; Higher scores indicate greater impairment in quality of life)
The effect of budesonide in functional dyspepsia on state of anxiety | At baseline, 8 weeks after start of treatment (9mg), 2 weeks after start of tapering (which is at 10 weeks), at the end of tapering (at 12 weeks), at 16 weeks (4 weeks after treatment discontinuation)
  The effect of budesonide in functional dyspepsia on state of anxiety, assessed by the Visceral Sensitivity Index (VSI) questionnaire (Likert scale from 1 to 6; 1 = not at all applicable, 6 = completely applicable; Score range: 15 (minimal sensitivity) to 90 (maximum sensitivity))
The effect of budesonide in functional dyspepsia on state of depression | At baseline, 8 weeks after start of treatment (9mg), 2 weeks after start of tapering (which is at 10 weeks), at the end of tapering (at 12 weeks), at 16 weeks (4 weeks after treatment discontinuation)
  The effect of budesonide in functional dyspepsia on state of depression, assessed by the Patient Health Questionnaire-9 (PHQ-9) questionnaire (9 questions, Likert scale 0-3; 0-4: Minimal or no depression; 20-27: Severe depression)
The effect of budesonide in functional dyspepsia on state of somatization | At baseline, 8 weeks after start of treatment (9mg), 2 weeks after start of tapering (which is at 10 weeks), at the end of tapering (at 12 weeks), at 16 weeks (4 weeks after treatment discontinuation)
  The effect of budesonide in functional dyspepsia on somatization, assessed by the PHQ 15 questionnaire (15 questions, Likert scale 0-2, 0 = Not bothered at all; 2 = Bothered a lot; score 0-4: Minimal somatization; score 15-30: High somatization)
The effect of budesonide in functional dyspepsia on barrier function by measuring mRNA levels of tight-junction related molecules | before treatment and 8 weeks after start of treatment (9 mg)
  The effect of budesonide in functional dyspepsia on mucosal permeability, including gene and protein expression of major tight-junction related molecules (Claudins, Occludin, ZO-1 (Zonula Occludens-1) by measuring mRNA levels using quantitative Polymerase Chain Reaction (qPCR) and Western Blot
The effect of budesonide in functional dyspepsia on barrier function by measuring mRNA levels of pro-inflammatory cytokines | before treatment and 8 weeks after start of treatment (9 mg)
  The effect of budesonide in functional dyspepsia on mucosal permeability, including gene and protein expression of pro-inflammatory cytokines by measuring mRNA levels using quantitative Polymerase Chain Reaction (qPCR) and Western Blot

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Yes
We are committed to ensuring transparency in our research. Individual Participant Data (IPD) will be made available upon reasonable request, provided it is necessary for publication in a peer-reviewed journal. Access will be granted in compliance with ethical guidelines and data protection regulations.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: During the peer-review process, Individual Participant Data (IPD) can be made available upon request to reviewers, provided it is necessary for the evaluation of the manuscript. After publication, IPD will also be accessible on a case-by-case basis, following a formal request and assessment to ensure compliance with ethical guidelines and data protection policies.
Access Criteria: Researchers interested in accessing the Individual Participant Data (IPD) are invited to contact the corresponding author directly.